CLINICAL TRIAL: NCT04020861
Title: Photobiomodulation Therapy and Transcutaneous Electrical Nerve Stimulation on Chronic Neck Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Richard Eloin Liebano, Professor, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 81711417.0.0000.5504
Record Dates: First submitted 2019-07-05; First posted 2019-07-16 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-06

CONDITIONS: Chronic Neck Pain
Keywords: Electrophysical agents; Low-level laser therapy; TENS; Neck pain; Chronic pain
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PBM + TENS (Active Comparator): The patients will be submitted to the active PBM and active TENS
  Interventions: Device: Active PBM; Device: Active TENS
- PBM (Active Comparator): The patients will be submitted to the active PBMT and placebo TENS
  Interventions: Device: Active PBM; Device: Placebo TENS
- TENS (Active Comparator): The patients will be submitted to the placebo PBMT and active TENS
  Interventions: Device: Active TENS; Device: Placebo PBM
- Placebo (Placebo Comparator): The patients will be submitted to the placebo PBMT and placebo TENS.
  Interventions: Device: Placebo PBM; Device: Placebo TENS

INTERVENTIONS:
Device: Active PBM — To active photobiomodulation therapy (PBMT) the patient will be oriented to lie preferably in prone. The treatment area will be defined according to painful area. In the active group will be used the followings parameters: low-level laser therapy, 808 nm, 4 infrared diodes, 180 mW, 9 J. In the placebo PBMT will be performed a simulation of laser application. The cluster probe will be positioned on painful area during the same time of active PBMT, the equipment will be turned on and set, however the trigger will be not actived and no beam will be applied.
  Arms: PBM; PBM + TENS
Device: Active TENS — To active transcutaneous electrical nerve stimulation (TENS) the patient will be oriented to lie preferably in prone. Two or four electrodes standard square self-adhesive electrodes (5 × 5 cm2) will be positioned according to the painful area related by patient. It will be used the following parameters: frequency of 100 Hz, pulse duration of 125 µs (positive phase), 30 minutes of current stimulation and the pulse amplitude will be increased until the patient reports a strong but comfortable paresthesia (including motor level stimulation but no painful TENS). The amplitude will be adjusted (if necessary) each 5 minutes to keep a strong but comfortable paresthesia.
  Arms: PBM + TENS; TENS
Device: Placebo PBM — In the placebo PBMT will be performed a simulation of laser application. The cluster probe will be positioned on painful area during the same time of active PBMT, the equipment will be turned on and set, however the trigger will be not actived and no beam will be applied.
  Arms: Placebo; TENS
Device: Placebo TENS — To placebo transcutaneous electrical nerve stimulation (TENS) Two or four electrodes standard square self-adhesive electrodes (5 × 5 cm2) will be positioned according to the painful area related by patient. This device was customized to deliver a current for 30 seconds (both channels) and then ramp off over the next 15 seconds so that it will be active for a total of 45 seconds. This will permit the patient to fell the TENS sensation while applying the settings.
  Arms: PBM; Placebo

SUMMARY:
This study evaluates the efficacy isolated and combinaded of photobiomodulation therapy with low level laser therapy and the transcutaneous electrical nerve stimulation.

DETAILED DESCRIPTION:
Non-specific chronic neck pain patients will be treated with low-level laser therapy and/or trancutaneous electricam nerve stimulation. They will receive 10 sessions of treatment. Before and after the treatment physical measures and psychosocial factors will be evaluted to verificy the efficay these electrophysical agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific chronic neck pain, defined as pain or discomfort in the posterior cervical region between the superior nuchal line and the first thoracic spinous process and / or shoulder girdle;
* Neck pain for at least 3 months;
* Neck Disability Index (NDI) score of 5 points or higher;
* Numeric Rating Scale (NRS) score of 3 or higher to pain intensity;
* Aged between 18 and 65 years;
* Men and women

Exclusion Criteria:

* Neck pain associated with nerve root compromise (measured by clinical examination of dermatomes, myotomes and reflexes);
* Previous spinal surgery;
* Patients treated with physical therapy for neck pain in the last 3 months previous the study;
* Severe spinal disorders such as fractures, tumors, inflammatory and infectious diseases;
* Any contraindication to low level laser therapy or transcutaneous electrical nerve stimulation;
* Rheumatic, metabolic, neurological or cardiopulmonary diseases;
* Patients who require artificial cardiac pacemakers;
* Skin diseases, mainly at the current application site;
* Tumors or cancer historic in the last 5 years;
* Pregnancy;
* If the patient started any physical activity in the last 2 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
Pain intensity: Numerical Rating Scale (Pain NRS) | 2 weeks after randomization
  Pain intensity will be evaluated using an 11-point (0-10) Numerical Rating Scale (Pain NRS), which is a simple and easy-to-use measuring scale that consists of a sequence of numbers from zero to 10, in which zero represents "no pain" and 10 represents "the worst pain imaginable". The pain evaluation will be carried out verbally with the patient reporting the pain intensity.

SECONDARY OUTCOMES:
Pain intensity: Numerical Rating Scale (Pain NRS) | 6 weeks after randomization
  Pain intensity will be evaluated using an 11-point (0-10) Numerical Rating Scale (Pain NRS), which is a simple and easy-to-use measuring scale that consists of a sequence of numbers from zero to 10, in which zero represents "no pain" and 10 represents "the worst pain imaginable". The pain evaluation will be carried out verbally with the patient reporting the pain intensity.
Pain intensity at movement: Numerical Rating Scale (Pain NRS) | 2 weeks after randomization
  Pain intensity will be evaluated during the cervical movements of flexion, extension, right and left lateral inclination and right and left rotation, using an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Neck disability | 2 weeks after randomization
  Neck disability will be evaluated using neck disability index (NDI) that consists of a 10-item questionnaire that assess the impact of pain on daily activities using a score from 0 to 5 for each section, with higher values indicating more severe impact.
Cervical range of motion | 2 weeks after randomization
  Cervical range of motion will be measured with a fleximeter
Pressure Pain Threshold | 2 weeks after randomization
  Pressure pain threshold (PPT) in the neck, shoulder girdle and anterior tibialis muscle will be measured using a Somedic Type II pressure algometer
Pain temporal summation (TS) | 2 weeks after randomization
  Temporal summation (TS) will be induced by a pressure algometer. Ten (10) stimuli with a pressure of 40 kPa/s of the mean value of algometry performed prior on the upper trapezius. Patients will be asked about their pain using NRS at the first, fifth and tenth stimulus.
Conditioned pain modulation (CPM) | 2 weeks after randomization
  The conditioned stimulus for eliciting CPM will be the cold pressor test (Cold Water Bath test to the hand) and the test stimulus will be the assessment of PPT on the upper trapezius muscle.
Depressive symptoms | 2 weeks after randomization
  The depressive symptoms will be performed using Beck Depression Inventory (BDI). The scale consists of items including symptoms and attitudes whose intensity range from neutral to a maximum level of severity, rated from 0 to 3.
Pain catastrophizing | 2 weeks after randomization
  Pain catastrophizing will be performed with Pain Catastrophizing Scale (PCS) - The PCS is a self-administered questionnaire that consists of 13 items to assess catastrophizers. The items are rated on a 5-point Likert-type scale in which both intensity and frequency information are represented, with the following ﬁve levels of response for each Likert item: (0) not at all, (1) to a slight degree, (3) to a moderate degree, (4) to a great degree, (5) and all the time. The total score is computed by summation of all items and the total score ranges from 0 to 52 points. Higher scores indicate greater catastrophic pain.
Change in patient perception of quality of life:12-Item Short-Form Health Survey (SF-12) | 2 weeks after randomization
  The quality of life will be performed using 12-Item Short-Form Health Survey (SF-12) version 2 questionnaire. This is a self-report measure that assesses physical (Physical Component Summary - PCS) and mental (Mental Component Summary - MCS) health on a scale of 0 - 100. Higher scores represent better levels of quality of life.
Analgesic intake | 2 weeks after randomization
  Anlgesic intake will be evaluated asking to the patients all analgesic medications (opioids and non-opioids) taken one week prior to evaluation and during the treatment.
Global perceived effect (GPE) | 2 weeks and 6 weeks after randomization
  Global perceived effect will be evaluated by an 11 - point (- 5 to + 5) Global Perceived Effect Scale. It consists of an 11-point scale that ranges from -5 (vastly worse) through 0 (no change) to 5 (completely recovered).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon requested of principal investigator.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Rampazo EP, de Andrade ALM, da Silva VR, Back CGN, Liebano RE. Photobiomodulation therapy and transcutaneous electrical nerve stimulation on chronic neck pain patients: Study protocol clinical trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Feb;99(8):e19191. doi: 10.1097/MD.0000000000019191. PMID 32080103